CLINICAL TRIAL: NCT04842071
Title: Open-label Clinical Trial on the Safety and Efficacy of 18F-sodium Fluoride (NaF) PET Imaging in Patients in Need of a Standard 99mTc Bone Scintigraphy
Brief Title: 18F-sodium Fluoride (NaF) PET to Replace Bone Scintigraphy: Safety and Efficacy Assessment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, Head of clinical research, CIMS, CRCHUS, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIMS-2008-01
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Bone Cancer; Articular Disease; Infectious Disease
Keywords: 18F-NaF; Bone scintigraphy; bone diseases
MeSH Terms: conditions — Bone Neoplasms; Joint Diseases; Communicable Diseases; Bone Diseases

STUDY DESIGN:
Intervention Model Description: Every patient in need and/or eligible for a standard 99mTc-biphosphonate bone scintigraphy is eligible to participate to this study. Patient data and examination results will be compiled and monitored. The safety profile of 18F-NaF produced in the primary site will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- 18F-NaF eligible patients (Experimental): Eligibility for 18F-NaF PET scans is the same than for bone scintigraphy routinely prescribed in the clinic.
  Interventions: Diagnostic Test: 18F-sodium fluoride

INTERVENTIONS:
Diagnostic Test: 18F-sodium fluoride — Intravenous injection of 4 MBq/kg for pediatric patients, or 5 MBq/kg for adult patients (maximum of 555 MBq), followed by a 45 minutes waiting time. Patients is then placed in supine position in a PET/CT scanner for a duration of no more than 30 minutes.
  Other Names: 18F-NaF

SUMMARY:
18F-sodium fluoride (18F-NaF) was already investigated numerous times in the last 40 years as a PET alternative to standard 99m-technetium-derived bone scintigraphy. However, lack of universal tracer availability and higher costs contributed to the failure of 18F-NaF to systematically supplant bone scintigraphy as a standard of care.

Recently, an isotope shortage crisis occurred and evidenced the need to have non-reactor-derived alternatives for many nuclear medicine procedures, including bone scintigraphy. Since 18F-NaF is cyclotron-produced, it could become a necessary alternative to bone scintigraphy in case of another worldwide isotope shortage.

The study aims to evaluate the safety profile of 18F-NaF injection. Moreover, a patient registry will be compiled in order to perform sub-studies on 18F-NaF diagnostic performance on diverse bone and articular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a 99mTc-biphosphonate bone scintigraphy is indicated;
* Pediatric patients for whom a 99mTc-biphosphonate bone scintigraphy is indicated for oncologic or infectious reasons
* Able to tolerate supine position
* Written consent

Exclusion Criteria:

* Healthy subjects
* Pregnancy
* Unable of maintaining supine position for more than 15 minutes
* Refusal to sign the consent form
* Known allergy or hypersensitivity to 18F-NaF or any of its constituants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety profile of 18F-NaF | 17 years
  A registry monitoring eventual adverse effects for this radiopharmaceutical agent will be compiled. Usual procedures will be applied to divulgate any serious adverse effects.
Efficacy profile of 18F-NaF compared to 99mTc-biphosphonate bone scintigraphy | 17 years
  Using the patient registry, and in the eventual sub-studies to come, the diagnostic performance of 18F-NaF-PET will be compared to similar available imaging tests, most notably 99mTc-biphosphonate bone scintigraphy.
Correlate 18F-NaF PET images with pathology reports | 17 years
  Pathology data from the diverse conditions eligible for the 18F-NaF PET scan will be also monitored when available. Prognostic value from the imaging data will be compared with those obtained from the pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Éric E Turcotte, MD, Principal Investigator — Université de Sherbrooke, Centre de Recherche du CHUS
Locations (2):
- Canada (2):
  - CHUS, Sherbrooke, Quebec
  - Université deSherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No